CLINICAL TRIAL: NCT05519033
Title: Pilondal Sinus Study: A National Survey
Brief Title: Pilonidal Sinus-Turkey
Acronym: PiSi
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Collaborators: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government); Ankara Oncology Research and Training Hospital (Network)
Responsible Party: Principal Investigator, Ali Yalcinkaya, MD, Gazi University
Other Study IDs: PISI-TR
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Pilonidal Sinus Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this research, main purpose is to determine the recurrence prevalence. Destination of the cohort study in which retroprospective data are prospectively reviewed, which aims to identify pilonidal disease subtypes for which various treatment options are indicated, identify various interventions, associate patients with the clinical stage, determine which results are meaningful to patients and which interventions they prefer and provide further research investigation recommendations. .

Primary outcome; To determine the postoperative recurrence rates according to the type of surgical intervention.

The secondary outcome is; to compare the overall patient satisfaction between different operative techniques and to obtain the ratio of different techniques applied for pilonidal sinus treatment in Turkey.

DETAILED DESCRIPTION:
In this study, the patient must be over 18 years of age for potential patient data for elective surgical treatment of pilonidal disease. The treatment techniques which considered eligible for the study should be determined by the surgical team and the patient information forms should be filled in at the hospital where the treatment was applied. Before collecting any patient data, the Lead Investigator or authorized research team member must be verified as suitable for the study.

Information should be processed on the Case Report Form (CRF) specifically designed for surgical intervention, and the surgeon's current practice should be in the information forms. Collected participant data will be recorded in the relevant CRFs and patient questionnaires. You should call to ask about the postoperative 1st day, 7th day, 6th month and 12th month status of the patients who provide the inclusion criteria and were operated during period -the defined by research protocol- . As a result; Since all patients who were operated between January 2019 and January 2020 and were included in the study completed their 12th month, the status of these patients in the specified dates will be questioned retrospectively and a prospective follow-up will not be performed. Later, the data will be transferred and entered into RedCAP, a remote web-based data collection system.

In CRF, the operations that the patient has had for pilonidal sinus treatment, the presence of postoperative recurrence, the time to return to normal activities, pain level and general treatment satisfaction are questioned.

ELIGIBILITY:
Inclusion Criteria:

- Symptomatic patient with the pilonidal sinus who is decided the treatment methods by the clinician.

Exclusion Criteria:

* Patients under 18 years of age asymptomatic (Stage I), acute abscess (Stage II), pregnant patients, presence of systemic disease such as DM, UC, Hidradenitis Suppurativa, patients with session hypersensitivity and the patients who are not authorized to give consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients ,with pilonidal sinus, treated by general surgeons
Sampling Method: Non-Probability Sample
Enrollment: 1742 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Postoperative Recurrence | 12 months
  Determine the postoperative recurrence rates according to type of surgical intervention.

SECONDARY OUTCOMES:
the ratio of different techniques methods | 12 months
  Compare the overall patient satisfaction between different operative techniques and to obtain the ratio of different techniques applied for pilonidal sinus treatment in Turkey.

CONTACTS AND LOCATIONS:
Overall Officials: Sezai Leventoglu, Proffesor, Study Chair — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)